CLINICAL TRIAL: NCT05150639
Title: Associations Between the Vaginal Microbiome, Inflammatory Status and Pregnancy Outcome - a Prospective, Observational Study in Women Undergoing Frozen Embryo Transfers.
Brief Title: Vaginal Microbiome and IVF Pregnancy Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Freya Biosciences ApS (Industry)
Collaborators: Boston IVF (Other)
Responsible Party: Sponsor
Other Study IDs: IVF-2
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Vaginal Flora Imbalance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples collected will be:
  Vaginal swabs Vaginal secretion Urine Menstrual effluent (optional) Peripheral blood (optional)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: IVF — Women planning to undergo frozen embryo transfer IVF procedure will be included. Samples will be obtained, but no study intervention will be applied. Pregnancy outcome data will be obtained, following frozen embryo transfer, to correlate against other data from samples (vaginal microbiome etc).

SUMMARY:
The aim of this prospective, observational study is to investigate the prevalence of vaginal dysbiosis among women undergoing IVF procedures in the US. And to investigate the associations between the vaginal microbiome and the pregnancy outcome following IVF.

DETAILED DESCRIPTION:
The present study will evaluate differences in vaginal microbiome composition in pregnant and non pregnant women who have undergone IVF treatment with frozen embryo transfer. Concurrently we aim to identify whether menstrual tissue and Cervicovaginal secretion possess complimentary biomarker information reflecting the immune/inflammatory status of the reproductive tract to determine its impact on pregnancy success following frozen embryo transfer IVF procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-44 years
* Patients whose written informed consent approved by the Institutional Review Board (IRB) has been obtained, after having been duly informed of the nature of the study and voluntarily accepted to participate after being fully aware of the potential risks, benefits and any discomfort involved.
* Women undergoing a planned frozen embryo transfer
* BMI between 18.5-35 kg/m2 (both included)
* Must be able to understand and read the informed consent form in English.

Exclusion Criteria:

* Current diagnosis of pathologies or malformations that affect the uterine cavity such as polyps, intramural myoma, adhesions, fibroids or hydrosalpinx.
* Any illness or medical condition that is unstable or which, according to medical criteria and Investigator's discretion may put at risk the patient's safety and her compliance in the study.
* Participants currently taking antibiotics or with any known condition requiring regular use of antibiotics, that would suggest the participant is likely to need antibiotic treatment during the observational period of this study.
* Systemic and/or vaginally applied antibiotic use within the last month prior to screening (except for prophylactic antibiotics related to egg retrieval).
* Patients utilizing oral contraceptive pills in the past month
* Latex or silicone allergy (Diva Cup and Vaginal Disc)

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women planning to undergo frozen embryo transfer IVF treatment at Boston IVF fertility clinic in Boston, US.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Prevalence of vaginal dysbiosis | Evaluated from sample collected 1 week prior to frozen embryo transfer
  The prevalence (evaluated as % of included population) of vaginal dysbiosis in women undergoing frozen embryo transfer IVF treatment in the US

SECONDARY OUTCOMES:
Associations of microbiome | Evaluated from sample collected 1 week prior to frozen embryo transfer and correlated with pregnancy outcomes obtained up until birth
  The difference in pregnancy success rates (biochemical pregnancy, clinical pregnancy and live birth) following frozen embryo transfer in women with versus without vaginal dysbiosis

CONTACTS AND LOCATIONS:
Overall Officials: Denis Vaughan, PhD, Principal Investigator — Boston IVF; Denny Sakkas, PhD, Principal Investigator — Boston IVF
Locations (1):
- Boston IVF The Waltham Center, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No